CLINICAL TRIAL: NCT02422095
Title: Registry of Endoscopic Ultrasound (EUS) Evaluation and Management of Pancreatic Fluid Collections and Pancreatic Cysts
Brief Title: Registry of Pancreatic Fluid Collections and Pancreatic Cysts
Status: Withdrawn | Type: Observational
Why Stopped: This is project was determined to be not research, and the IRB has no oversight
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 700323; 1108594 (Registry Identifier: Registry of Pancreatic Fluid Collections)
Record Dates: First submitted 2015-02-23; First posted 2015-04-21 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Fluid Collections; Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pancreatic fluid collections: Patients with pancreatic fluid collections undergoing endoscopy-based (EUS-guided) interventions
  Interventions: Procedure: Endoscopy-based (EUS-guided) interventions for pancreatic fluid collections
- Pancreatic cysts: Patients with pancreatic cysts undergoing EUS examination and possible EUS-guided sampling of cystic fluid.
  Interventions: Procedure: EUS of pancreatic cysts

INTERVENTIONS:
Procedure: Endoscopy-based (EUS-guided) interventions for pancreatic fluid collections — Data included are patient demographics, symptoms, disease severity, procedural indications, details of the pancreatic fluid collection on cross-sectional imaging/EUS, review of laboratory results/imaging, details of interventions, clinical response to intervention, adverse events from interventions and pancreatitis/pancreatic fluid collections, response to treatment including any recurrent hospital admissions, recurrence of pancreatic fluid collections, need for repeat interventions, details of pancreatic duct integrity (e.g. presence of disconnected pancreatic duct syndrome), and clinical status at follow-up.
  Groups: Pancreatic fluid collections
Procedure: EUS of pancreatic cysts — Data included are patient demographics (age, gender, race), symptoms at presentation, imaging modality performed to detect the cyst, cyst features on EUS, technical details of EUS-guided sampling, results of cyst fluid analysis, final diagnosis, any follow up and repeat examinations and details of any treatment performed.
  Groups: Pancreatic cysts

SUMMARY:
This registry aims to assess the outcomes of patients undergoing EUS-guided interventions of pancreatic fluid collections and EUS examination of pancreatic cyst lesions.

DETAILED DESCRIPTION:
For pancreatic fluid collections, data included in this registry are 292 variables on patient demographics (age, gender, race), symptoms at presentation, severity of disease prior to intervention, indications for undergoing endoscopic intervention, details of the pancreatic fluid collections on cross-sectional imaging and EUS, review of laboratory results, review of imaging, details of interventions performed for pancreatic fluid collections, clinical details following intervention, adverse events from interventions and pancreatitis/pancreatic fluid collections, interventions for any adverse events, response to treatment of pancreatic fluid collections including any hospital readmissions, recurrence of pancreatic fluid collections, need for repeat interventions for pancreatic fluid collections, details of pancreatic duct integrity such as the presence of disconnected pancreatic duct syndrome, and clinical status at follow-up.

For pancreatic cysts, data included in this registry are 60 variables on patient demographics (age, gender, race), symptoms at presentation, imaging modality performed to detect the cyst, features of the cyst on EUS, features of the main pancreatic duct on EUS, technical details of EUS-guided sampling of the cystic fluid, results of cyst fluid analysis including cytology, tumor markers, amylase levels, molecular markers, final diagnosis of the cyst on follow-up, details of any follow up evaluation performed, details of repeat examinations performed and details of any treatment performed for the pancreatic cyst.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 18 years or over, who are undergoing EUS evaluation of a pancreatic cyst lesion or endoscopy-based (EUS-guided) interventions for pancreatic fluid collection at the Center for Interventional Endoscopy will be included in this registry.

Exclusion Criteria

1. Age less than 18 years
2. No pancreatic cyst on EUS examination or no pancreatic fluid collection amenable to endoscopic drainage on EUS examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or over undergoing EUS evaluation of pancreatic cyst lesions or endoscopy-based (EUS-guided) interventions of pancreatic fluid collections.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success in patients with pancreatic fluid collections following endoscopic interventions | 6 months (minimum)
  The treatment success of a structured, algorithmic approach to the management of pancreatic fluid collections will be evaluated. Structured approach involves management strategies based on the type (pseudocyst vs. necrosis), size, number, location of the pancreatic fluid collection, degree of necrosis, need for adjunctive percutaneous drain placement, and presence of disconnected pancreatic duct syndrome.
Natural history and disease progression in pancreatic cysts | 6 months (minimum) to 5 years
  The relationship between patient characteristics, clinical symptoms, cyst and pancreatic duct characteristics on cross-sectional imaging and on EUS examination, results of cyst sampling (including cytology, tumor markers, amylase, molecular markers) and final diagnosis on follow-up with be determined.

SECONDARY OUTCOMES:
Number of interventions required for treatment success in patients with pancreatic fluid collections | 6 months (minimum)
  The total number of procedures (including transmural drainage and endoscopic necrosectomy) required to achieve treatment success (defined as resolution of symptoms and fluid collection on imaging) in patients with pancreatic fluid collections at 6 months follow up.
Treatment failure in patients with pancreatic fluid collections | 6 months (minimum) to 5 years
  The rate of failure (defined as need for rescue surgery or death due to underlying disease or intervention) of EUS-guided treatment of pancreatic fluid collections will be assessed
Adverse events in patients undergoing EUS-guided drainage of pancreatic fluid collections | 6 months (minimum) to 5 years
  The rate and type of adverse events in patients undergoing EUS-guided drainage of pancreatic fluid collections will be assessed
Impact of disconnected pancreatic duct syndrome in patients undergoing EUS-guided drainage of pancreatic fluid collections | 6 months (minimum) to 5 years
  The impact of disconnected pancreatic duct syndrome in patients undergoing EUS-guided drainage of pancreatic fluid collections on treatment success and disease recurrence will be assessed.
Impact of placement of long-term plastic transmural stents in patients with pancreatic fluid collections and disconnected pancreatic duct syndrome | 6 months (minimum) to 5 years
  The impact of placement of long-term plastic transmural stents in patients with pancreatic fluid collections and disconnected pancreatic duct syndrome will be assessed.
Treatment success in patients with pancreatic fluid collections undergoing a structured approach to endoscopic necrosectomy following EUS-guided drainage of pancreatic fluid collections | 6 months (minimum) to 5 years
  The treatment success of a structured approach endoscopic necrosectomy following EUS-guided drainage of pancreatic fluid collections will be assessed. The structured approach to endoscopic necrosectomy involves three steps - debridement, extraction and irrigation.
Hospital admissions and reinterventions in patients undergoing EUS-guided drainage of pancreatic fluid collections | 6 months (minimum) to 5 years
  The number of hospital admissions and reinterventions in patients undergoing EUS-guided drainage of pancreatic fluid collections will be assessed
Recurrence of pancreatic fluid collections in patients undergoing EUS-guided drainage of pancreatic fluid collections | 6 months (minimum) to 5 years
  The rate of recurrence of pancreatic fluid collections in patients undergoing EUS-guided drainage of pancreatic fluid collections will be assessed
Evaluate the role of plastic stents in patients undergoing EUS-guided drainage of pancreatic fluid collections. | 6 months (minimum) to 5 years
  Evaluate the role of plastic stents in the era of LAMS specifically pertaining to a) exchange of LAMS for plastic stents in patients with disconnected pancreatic duct syndrome after PFC resolution and b) use of plastic stents as the primary mode of drainage in patients with pseudocysts and obstructive/disconnecte main pancreatic duct.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — Florida Hospital Center for Interventional Endoscopy
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript will be developed following study closure.

REFERENCES:
- [Derived] Bang JY, Mel Wilcox C, Arnoletti JP, Varadarajulu S. Importance of Disconnected Pancreatic Duct Syndrome in Recurrence of Pancreatic Fluid Collections Initially Drained Using Lumen-Apposing Metal Stents. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1275-1281.e2. doi: 10.1016/j.cgh.2020.07.022. Epub 2020 Jul 16. PMID 32683101
- [Derived] Bang JY, Hawes RH, Varadarajulu S. Lumen-apposing metal stent placement for drainage of pancreatic fluid collections: predictors of adverse events. Gut. 2020 Aug;69(8):1379-1381. doi: 10.1136/gutjnl-2019-320539. Epub 2020 Feb 17. No abstract available. PMID 32066622